CLINICAL TRIAL: NCT06212349
Title: Effect of a Therapeutic-educational Physiotherapy Program on Pain and the Physical-functional Sphere in Women With Endometriosis and Its Impact on Quality of Life
Brief Title: Therapeutic-educational Physiotherapy on Pain, Physical-functionality and Quality of Life in Women With Endometriosis.
Acronym: PHYSIO_ENDOM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Hospital Universitario La Fe (Other); Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Principal Investigator, Laura Fuentes Aparicio, Doctor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UV_Dep_FISIO
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Endometriosis; Chronic Pain; Women's Health
Keywords: endometriosis; Chronic Pain; Physical Therapy; Health education; Women
MeSH Terms: conditions — Endometriosis; Chronic Pain; Health Education

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): They will receive therapeutic-educational physiotherapy, which will combine therapeutic exercise with a pain education program,
  Interventions: Other: therapeutic-educational physiotherapy and pain education program
- Control (Other): They will receive the pain education program.
  Interventions: Other: pain education program

INTERVENTIONS:
Other: therapeutic-educational physiotherapy and pain education program — The EG will carry out a total of 24 sessions, at a rate of 3 weekly sessions of 30 minutes each. The first session of each month will be in person and the rest will be done at home following video tutorials with an App (https://fisiotrack.com). The face-to-face sessions will be conducted by a women's health physiotherapist, and will consist on therapeutic exercises based on body awareness, motor control and respiratory awareness.They will also receive a pain education program with indications on pain education, as well as basic information and general advice on the positive effects of physical activity and a healthy lifestyle for endometriosis. In addition, biweekly supervision will be carried out via telephone or video conference by a specialized physiotherapist.
  Arms: Experimental
Other: pain education program — They will receive instructions on pain education, as well as basic information and general advice about the positive effects of physical activity and a healthy lifestyle for your endometriosis, in writing via email. In addition, they will receive biweekly supervision via telephone or video conference by a specialized physical therapist.
  Arms: Control

SUMMARY:
This is a randomized clinical trial that will be carried out in women with endometriosis divided into two groups: the experimental group (EG) that will receive therapeutic-educational physiotherapy, which will combine therapeutic exercise with a pain education program, and the control group (CG) who will receive the pain education program.

The participants will be evaluated at three moments: before starting the study (T1), after the 8-week treatment program (T2) and after another 8 weeks of follow-up in which they will be encouraged to continue with the treatment (T3). The initial assessment will include a medical and physiotherapy history, and at T1, T2 and T3 the following will be assessed: pain, abdominopelvic mobility, muscle status, functionality, sexual function, quality of life, stress and biomarkers of chronic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of endometriosis made by imaging techniques (MRI or ultrasound) or by surgery.
* A period of 3 months or more since the last surgery if they have undergone surgery.
* Who are receiving hormone treatment and have their disease under control.
* Persistent pelvic pain for at least 3 months.
* With pain and hypertonus in the pelvic musculature, myofascial syndrome, vestibulodynia or pudendal neuropathy.
* Consent to participate in the study
* Capable of carrying out the follow-up of the study until the final visit.
* Who have audiovisual resources and the internet at their disposal.

Exclusion Criteria:

* Women in the menopausal phase
* Women undergoing fertility treatment or planning to undergo fertility treatment in the next 3 months.
* Pregnant women.
* Women undergoing physiotherapy treatment or who have undergone physiotherapy treatment in the last 3 months.
* Having suffered a fracture in the last 3 months in the lower limb that limits their functional capacity.
* Cognitive illness that prevents correct comprehension of the exercises.
* Musculoskeletal pathology or neuropathy in acute phase.
* Having suffered or suffering from a neoplastic disease.
* Untreated endometriosis
* Acquired genital abnormalities of the pelvis or pelvic floor.
* Women in a situation of litigation or economic compensation, or pending the granting of a degree of disability.
* Severe mental illness (schizophrenia, borderline personality disorder, etc.)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 62 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2024-12-14 (Actual); Study Completion 2026-12-22 (Estimated)

PRIMARY OUTCOMES:
Musculoskeletal pain - Pressure pain threshold | 3 assessent times: T1(pre-intervention), T2 (after 8 weeks intervention), T3 (after 16 weeks intervention)
  Pressure pain threshold measured in rectus abdominis and lumbar muscles
Musculoskeletal pain - quantitative Sensory Testing | 3 assessent times: T1(pre-intervention), T2 (after 8 weeks intervention), T3 (after 16 weeks intervention)
  Quantitative sensory testing is a non-invasive technique used to assess and quantify sensory functions by determining sensation and pain thresholds using pressure.
Musculoskeletal pain - pain drawing | 3 assessent times: T1(pre-intervention), T2 (after 8 weeks intervention), T3 (after 16 weeks intervention)
  Identification of pain areas through a pain map: this consists of a human figure on a two-dimensional plane on which the patient can express the representation of the pain areas on a schematic of the body surface.
Musculoskeletal pain - Central Sensitisation Inventory | 3 assessent times: T1(pre-intervention), T2 (after 8 weeks intervention), T3 (after 16 weeks intervention)
  Central Sensitisation Inventory: is a self-report instrument that indirectly assesses somatic and emotional symptoms that have been found to be associated with Central Sensitisation.

SECONDARY OUTCOMES:
Physical-Funcionality - Hand grip Strength | 3 assessent times: T1(pre-intervention), T2 (after 8 weeks intervention), T3 (after 16 weeks intervention)
  Hand grip strength will be measured by the handgrip strength technique using a Jamar Plus+ digital hand dynamometer.
Physical-Funcionality - functional performance | 3 assessent times: T1(pre-intervention), T2 (after 8 weeks intervention), T3 (after 16 weeks intervention)
  To assess functional performance patients will be instructed to cross their arms over their chest and complete as many standing cycles as possible in 30 s (30 second- Sit to stand).
Physical-Funcionality- Pelvic floor Dynamometry | 3 assessent times: T1(pre-intervention), T2 (after 8 weeks intervention), T3 (after 16 weeks intervention)
  Dynamometry of the pelvic floor muscles: measurement of basal tone (g) and tone at maximum contraction (Phenix Liberty Dynamometer).
Physical-Funcionality - Body composition | 3 assessent times: T1(pre-intervention), T2 (after 8 weeks intervention), T3 (after 16 weeks intervention)
  Body composition (% fat, % water, % muscle): record body composition (skeletal muscle mass and % body fat) with a bioimpedance scale (DC-430MA, Tanita Corporation of America, Inc, Arlignton Heights, IL, USA).
Physical-Funcionality - Motor control | assessent times: T1(pre-intervention), T2 (after 8 weeks intervention), T3 (after 16 weeks intervention)
  Determine motor control: clinical test of lumpopelvic and thoracolumbar dissociation will be used.
Physical-Funcionality - Lumbar spine flexibility | assessent times: T1(pre-intervention), T2 (after 8 weeks intervention), T3 (after 16 weeks intervention)
  Lumbar spine flexibility: It will be measured with the Schöber test
Physical-Funcionality - Catastrophyzing | assessent times: T1(pre-intervention), T2 (after 8 weeks intervention), T3 (after 16 weeks intervention)
  Catastrophyzing: to assess catastrophic thinking related to pain the Pain Catastrophyzing Scale (PCS) will be used
Physical-Funcionality - Kinesophobia | assessent times: T1(pre-intervention), T2 (after 8 weeks intervention), T3 (after 16 weeks intervention)
  Kinesophobia: it will be assessed with the Tampa Scale for Kinesophobia-11 (TSK-11), which consists of 11 items.
Quality of Life - Endometriosis | assessent times: T1(pre-intervention), T2 (after 8 weeks intervention), T3 (after 16 weeks intervention)
  Quality of life will be assessed using the Spanish version of the Endometriosis Health Profile-30 (EHP-30).
Quality of Life - Gastrointestinal | assessent times: T1(pre-intervention), T2 (after 8 weeks intervention), T3 (after 16 weeks intervention)
  Quality of life at the gastrointestinal level will be assessed using the Gastrointestinal Quality of Life Index, which addresses 5 domains (digestive symptoms, physical state, emotions, social dysfunction and effects of medical treatment).
Quality of Life - Sexual Function | assessent times: T1(pre-intervention), T2 (after 8 weeks intervention), T3 (after 16 weeks intervention)
  the abbreviated Index of Female Sexual Function (IFSF-6) will be used. It is a multidimensional self-reported instrument for the evaluation of female sexual function
Quality of Life - Stress | assessent times: T1(pre-intervention), T2 (after 8 weeks intervention), T3 (after 16 weeks intervention)
  Stress using the Perceived stress scale (PSQ).
Biomarkers - Inflamation | assessent times: T1(pre-intervention), T2 (after 8 weeks intervention), T3 (after 16 weeks intervention)
  Plasma markers of chronic inflammation and intestinal permeability will be assessed including a multiplex array of inflammation markers, and as specific markers of chronic inflammation associated with intestinal permeability, zonulin, C-reactive protein, Binding Protein , and bactericidal/permeability-increasing protein will be assessed.
Patient's satisfaction | assessent times: T2 (after 8 weeks intervention), T3 (after 16 weeks intervention)
  Satisfaction with the treatment received will be assessed using the Satisfaction with Treatment Received Scale (CRES-4).
Patient's perception of change | assessent times: T2 (after 8 weeks intervention), T3 (after 16 weeks intervention)
  Patient's Perception of change after the treatment will be measured by patients' global impression of change (PGIC) in a quantitative and qualitative way.
APP usability | assessent times: T2 (after 8 weeks intervention), T3 (after 16 weeks intervention)
  A questionnaire on the usability of the application will be used. System Usability Scale.
Adherence to treatment | assessent times: T2 (after 8 weeks intervention), T3 (after 16 weeks intervention)
  Adherence to treatment: in the experimental group it will be measured through the records made in the application https://fisiotrack.com/, in the control group it will be measured through an ad hoc activity diary that will be provided to them.

CONTACTS AND LOCATIONS:
Overall Officials: laura Fuentes Aparicio, PhD, Principal Investigator — University of Valencia
Locations (1):
- Hospital Universitari i Politècnic La Fe,, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No